

## **Consent form**

Glycaemic Response (GR), Insulin Response (IR), glucagon-like peptide-1 (GLP-1) and gastric inhibitory polypeptide (GIP) response study

## Contacts:

Dr. Helen Lightowler, Director of the Oxford Brookes Centre for Nutrition and Health

Dr. Sangeetha Thondre, Senior Lecturer in Nutrition

Oxford Brookes Centre for Nutrition and Health Department of Sport and Health Sciences Faculty of Health and Life Sciences Oxford Brookes University Gipsy Lane Campus Oxford OX3 0BP

Tel: 01865 484365/ 01865 483988/

Email: hlightowler@brookes.ac.uk / Pthondre@brookes.ac.uk

| Ρle | ease <u>INITIAL</u> the appropriate box | | |
|---|---|---|---|
| | | Yes | No |
| 1. | I confirm that I have read and understand the information sheet for the above research project. | | |
| 2. | I confirm that I have had the opportunity to ask questions and have received satisfactory answers to all my questions. | | |
| 3. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving reason, or to withdraw any unprocessed data previously supplied. | | |
| 4. | I understand that confidentiality of information provided can only be protected within the limits of the law. | | |
| 5. | I agree to take part in the above research. | | |
| | me of Participantock capitals) | Date | |
| Się | gnatureConta | act number: | |
| en | nail: | | |
| Na | me of Researcher | | |
| (bl | ock capitals) | | |
| Się | nature | | |
| This project is funded by Roquette Frères 27 <sup>tl</sup> | | <sup>th</sup> Novembe | r 2018 |